CLINICAL TRIAL: NCT04794504
Title: Botulinum Toxin Type A Injected Into the Temporalis and Masseter Before Orthognathic Surgery to Improve Postoperative Pain
Brief Title: Investigating Temporalis and Masseter Botox Injection Before Orthognathic Surgery to Improve Postoperative Pain
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kingsway Oral & Maxillofacial Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CCF2021; 248417 (Other: Health Canada)
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Intervention Model Description: We will have two independent groups, one receiving botox injection, and another receiving saline injection.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All sponsors and collaborators will be blinded, and randomization and mixing of solutions will be done by an assistant not involved in the study. Half way through the study, one of the members of the research team will be unblinded to ensure confounders are appropriately matched in each of the two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botox Injection Group (Experimental): Two weeks pre-operatively, patients in the Botox injection group will receive intramuscular injections of Botox totaling 100U bilaterally (50U/side). 10 U will be injected into the temporalis (over 5 sites) and 40 U will be injected into the masseter muscle (over 4 sites). Botox will be reconstituted from a powdered form in 2cc of 0.9% sterile saline, and appropriate volumes will be administered.
  Interventions: Drug: Botox 100 UNT Injection
- Saline Injection Group (Placebo Comparator): Two weeks pre-operatively, patients in the saline injection group will receive intramuscular injections of Botox totaling the same volumes administered for Botox patients above, across the same number of sites in the temporalis and masseter muscles bilaterally.
  Interventions: Other: 0.9% Saline Injection

INTERVENTIONS:
Drug: Botox 100 UNT Injection — Botox will be injected intramuscularly into the masseter and temporalis muscles bilaterally to investigate if it can supplement postoperative analgesia in orthognathic surgery patients
  Other Names: OnabotulinumtoxinA
  Arms: Botox Injection Group
Other: 0.9% Saline Injection — As a placebo control to the 100 UNT Botox injection, 0.9% saline will be injected intramuscularly into the masseter and temporalis muscles bilaterally
  Arms: Saline Injection Group

SUMMARY:
Jaw surgery has become a very successful way to improve the appearance and functional needs of patients. Like any surgery, jaw surgery comes with a host of possible issues that patients may experience during their recovery. Although some of the most serious complications, like infections, have reliable ways to alleviate the symptoms, patients must endure several other discomforting factors. These include postoperative pain and muscle spasms. Botox® is becoming an increasingly used intervention to treat muscle related disorders (including temporomandibular disorders and chronic myofascial pain) in the head and beck region. The investigators believe that by injecting Botox® into the muscles surrounding the surgical area, patients may experience a relief in tension-related discomfort, leading to less pain and better jaw function during recovery from surgery. Further, the side effects of Botox® are either very minimal or exceedingly rare. Ultimately, Botox® may serve as a great alleviating factor with few downsides, and represent a supplementary approach to helping mitigate postoperative pain.

DETAILED DESCRIPTION:
Background and Rationale: Dentofacial deformities in the maxillofacial skeleton often require surgical intervention to correct aesthetic and functional deficiencies (Naran, Steinbacher, and Taylor, 2018). Often, patients suffer a number of postoperative complications, including postoperative pain and muscle spasms (Phillips, Blakey, and Jaskolka, 2008). While post-operative analgesics are used, regimens are often unsatisfactory in their ability to alleviate patient discomfort (Raschke et al. 2018). Botulinum toxin type A variants (BoNT-A; including Botox®) are becoming an increasingly used intervention to treat muscle-related disorders in the head and neck region, including migraines, myofascial pain, and temporomandibular joint disorders (Walker & Dayan, 2014; Dodick et al, 2010; Mimeh, Fenech, Myers, & Ghanem, 2019; Khalifeh et al., 2016, Machado et al., 2020). This occurs by inducing a flaccid muscle paralysis, which alleviates tension-related discomfort (Kwon et al., 2019). Thus by injecting Botox® into the muscles surrounding the surgical area preoperatively, patients may experience a relief in tension-related muscle pain and better jaw function during recovery from surgery. In addition to its great safety profile, where side effects are either very minimal or exceedingly rare, Botox® may serve as a great supplemental option to current postoperative analgesic regimens (Dressler et al., 2015, Yeh et al., 2018).

Objective: The primary objective of this study is to investigate whether preoperative injection of Botox® into the temporalis and masseter in patients undergoing bilateral sagittal split osteotomies (BSSO) will improve pain scores and spasms in the immediate 2 week, as well as 6 week, postoperative periods. Additionally, patients will be followed 5 years from the time of surgery to look for indicators of relapse, including infection and hardware failure.

Research question: Can injecting Botox® into facial muscles 2 weeks prior to orthognathic surgery result in decreased pain and muscle spasms postoperatively?

Methods: The investigators plan to do a pilot study involving patients undergoing BSSO to evaluate postoperative pain scores and muscle spasms. There is a lack of evidence investigating post-operative pain management in orthognathic surgery using Botox®, thus the studies outlined in this proposal will serve as a pilot project. However, to guide sample size determination, another study investigating incobotulinumtoxinA, one of the variants of botulinum toxin with a similar potency profile to Botox® (Scaglione, 2016), was used. This product has been used as a therapeutic treatment for temporomandibular disorders to manage myofascial pain (Patel, Lerner, and Blitzer, 2017). For these studies, based on previous experiences, a pain difference of 15% was determined to be clinically significant. Assuming a normal distribution, a continuous pain outcome, with an ⍺-level of 0.05, and a power of 80%, the investigators estimate 32 patients/group will need to be enrolled to capture this difference.

This will be a double-blinded study. The patients, principal investigators and trained observers analyzing the data will be blinded to the two groups. Half of the patients will receive BoNT-A injections (Botox® Therapeutic by Allergan, Inc), with the other half receiving 0.9% normal saline injections as a control cohort. Injections for both cohorts will be done two weeks preoperatively. Patients will be randomly designated to one of the two groups by a research assistant at Kingsway Oral and Maxillofacial surgery not named to the investigative team. Patients will be randomized into two groups using a 2:2 randomized block design. A computer-generated algorithm developed the randomization sequence which allowed for allotment of each patient into either group 1 (indicating Botox® injection) or 2 (indicating saline injection). Patients will not be informed of the group they belong to, only that they will be injected with either Botox® or saline; the surgical assistants will prepare either the Botox® injection or the 0.9% normal saline injection. The injection will be given to the surgeons performing the procedures with no knowledge of which patients will be getting which injection.

BSSO will be performed by Dr. Clayton Davis, Dr. Kevin Lung, and Dr. Matt Fay according to Kinsgway Oral and Maxillofacial Surgery clinical protocols. Patients will be asked to complete a numerical response scale (NRS) daily for 14 consecutive days, starting on postoperative day 1. Each day, the highest pain rating will be recorded as a whole number on a 0-10 scale. In the same 2 week timeframe, patients will also be asked to track any muscle spasms daily in the form of a "yes/no" question. At the 6 week follow-up appointment, patients will be asked to rate their pain at the current time on the NRS, and will be asked about further muscle spasms in the 2-6 week postoperative period in the form of a "yes/no" question. In order to track pain scores and muscle spasms, a paper questionnaire will be distributed to all patients. In addition to scoring pain daily on the NRS, patients will be asked to track: the time of the most severe pain, medications that were taken to help with the pain, pain intensity 1 hour after medication was taken, location of the pain, activities that led to onset of pain, and occurrence of muscle spasms. At the 2 week follow-up appointment, patients will bring back their paper copy of the questionnaire. Hardware failure and infection will be documented in the patient's chart, and will be viewed retrospectively study 5 years from now in the form of chart reviews of all study participants.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages 18 and 65 undergoing BSSO at Kingsway Oral and Maxillofacial Surgery are eligible to participate in the study, provided they do not fit any of the exclusion criteria.

Exclusion Criteria:

-Patient with history of chronic pain conditions including, but not limited to: myofascial pain:

* TMD, internal disc derangement, and TMJ osteoarthritis
* chronic migraines/tension type headaches and cervical pain
* generalized anxiety disorder
* diagnosed neuropathic pain (neuralgias)
* Mentally incompetent individuals
* History of botulinum toxin use for cosmetic and therapeutic uses
* History of trauma or previous orthognathic surgery
* Patients with hypersensitivity to BoNT-A
* Pregnant women
* Nursing women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-04-19 (Estimated); Primary Completion 2022-04-19 (Estimated); Study Completion 2026-04-19 (Estimated)

PRIMARY OUTCOMES:
Investigating a role of Botox intramuscular injection in reducing postoperative pain scores in orthognathic surgery patients 2 and 6 weeks after surgery | Analysis of this outcome will be ongoing throughout the study duration, and will end with the final orthognathic surgery patient completing their 2 week pain assessment
  At a two week endpoint postoperatively, orthognathic surgery patients will be asked to submit the results of the 2-week numerical rating scale questionnaire. The numerical rating scale will be administered from 0 to 10 (integer values only), with 0 representing no pain, and 10 representing the most severe pain. Co-investigators will gather this data, and the blinding protocol will be broken after the final participant submits their questionnaire to assign patients into their appropriate groups for analysis. Pain score trends between the Botox® and saline groups will be compared on a day-to-day basis, with potential use of area under curve analysis to get a scope of the overall pain scores over the 14 day postoperative period. Single pain scores at a 6 week follow-up appointment will also be collected.

SECONDARY OUTCOMES:
Investigating a role of Botox intramuscular injection in reducing postoperative muscle spams orthognathic surgery patients 2 weeks after surgery | Analysis of this outcome will be ongoing throughout the study duration, and will end with the final orthognathic surgery patient completing their 6 week pain assessment
  At the 6 week follow-up appointment, patients will be asked if they experienced muscle spasms in the 2-6 week postoperative period. Answers will be collected and reported as a proportion answering "yes" and "no", comparing the botox injection and saline injection groups
Investigating a role of Botox intramuscular injection in reducing hardware failure and rates of infection 5 years postoperatively | Analysis of this outcome will be ongoing throughout the study duration, and will end 5 years from the final participants day of surgery
  Five years after initiating this study, a retrospective analysis will be performed of participant's chart to note any infections or hardware failures that occurred, and if differences between the botox injection and saline injection group exist in these parameters
Investigating a role of Botox intramuscular injection in reducing postoperative pain scores in orthognathic surgery patients 6 weeks after surgery | Analysis of this outcome will be ongoing throughout the study duration, and will end with the final orthognathic surgery patient completing their 6 week pain assessment
  Single pain scores on a 0-10 numerical rating scale will be collected at a 6 week follow-up appointment with 0 representing no pain, and 10 being the most severe pain.

IPD SHARING:
Plan to Share IPD: No
IPD will be kept strictly confidential to the sponsors and scientific team appointed to this study by HREBA, and will not be distributed to other researchers.

REFERENCES:
- [Background] Scaglione F. Conversion Ratio between Botox(R), Dysport(R), and Xeomin(R) in Clinical Practice. Toxins (Basel). 2016 Mar 4;8(3):65. doi: 10.3390/toxins8030065. PMID 26959061
- [Background] Patel AA, Lerner MZ, Blitzer A. IncobotulinumtoxinA Injection for Temporomandibular Joint Disorder. Ann Otol Rhinol Laryngol. 2017 Apr;126(4):328-333. doi: 10.1177/0003489417693013. Epub 2017 Feb 1. PMID 28290229
- [Background] Naran S, Steinbacher DM, Taylor JA. Current Concepts in Orthognathic Surgery. Plast Reconstr Surg. 2018 Jun;141(6):925e-936e. doi: 10.1097/PRS.0000000000004438. PMID 29794714
- [Background] Phillips C, Blakey G 3rd, Jaskolka M. Recovery after orthognathic surgery: short-term health-related quality of life outcomes. J Oral Maxillofac Surg. 2008 Oct;66(10):2110-5. doi: 10.1016/j.joms.2008.06.080. PMID 18848110
- [Background] Raschke GF, Meissner W, Peisker A, Djedovic G, Rieger U, Guentsch A, Dammeier MG, Schultze-Mosgau S. Bilateral sagittal split osteotomy-parameters and correlations of postoperative pain management. Clin Oral Investig. 2018 Jan;22(1):181-187. doi: 10.1007/s00784-017-2097-z. Epub 2017 Mar 14. PMID 28293792
- [Background] Walker TJ, Dayan SH. Comparison and overview of currently available neurotoxins. J Clin Aesthet Dermatol. 2014 Feb;7(2):31-9. PMID 24587850
- [Background] Dodick DW, Turkel CC, DeGryse RE, Aurora SK, Silberstein SD, Lipton RB, Diener HC, Brin MF; PREEMPT Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: pooled results from the double-blind, randomized, placebo-controlled phases of the PREEMPT clinical program. Headache. 2010 Jun;50(6):921-36. doi: 10.1111/j.1526-4610.2010.01678.x. Epub 2010 May 7. PMID 20487038
- [Background] Kwon KH, Shin KS, Yeon SH, Kwon DG. Application of botulinum toxin in maxillofacial field: part I. Bruxism and square jaw. Maxillofac Plast Reconstr Surg. 2019 Oct 1;41(1):38. doi: 10.1186/s40902-019-0218-0. eCollection 2019 Dec. PMID 31649901
- [Background] Mimeh H, Fenech Magrin AM, Myers S, Ghanem AM. A Critical Review of Botulinum Toxin Type A in the Prophylactic Treatment of Chronic Migraine in Adults. Aesthet Surg J. 2019 Jul 12;39(8):898-907. doi: 10.1093/asj/sjy224. PMID 30184084
- [Background] Khalifeh M, Mehta K, Varguise N, Suarez-Durall P, Enciso R. Botulinum toxin type A for the treatment of head and neck chronic myofascial pain syndrome: A systematic review and meta-analysis. J Am Dent Assoc. 2016 Dec;147(12):959-973.e1. doi: 10.1016/j.adaj.2016.08.022. Epub 2016 Oct 10. PMID 27737756
- [Background] Machado D, Martimbianco ALC, Bussadori SK, Pacheco RL, Riera R, Santos EM. Botulinum Toxin Type A for Painful Temporomandibular Disorders: Systematic Review and Meta-Analysis. J Pain. 2020 Mar-Apr;21(3-4):281-293. doi: 10.1016/j.jpain.2019.08.011. Epub 2019 Sep 9. PMID 31513934
- [Background] Dressler D, Saberi FA, Kollewe K, Schrader C. Safety aspects of incobotulinumtoxinA high-dose therapy. J Neural Transm (Vienna). 2015 Feb;122(2):327-33. doi: 10.1007/s00702-014-1252-9. Epub 2014 Jul 17. PMID 25030362
- [Background] Yeh YT, Peng JH, Peng HP. Literature review of the adverse events associated with botulinum toxin injection for the masseter muscle hypertrophy. J Cosmet Dermatol. 2018 Oct;17(5):675-687. doi: 10.1111/jocd.12721. Epub 2018 Aug 9. PMID 30091170